CLINICAL TRIAL: NCT02447965
Title: Pilot Study: Rectus Sheath Blocks for Improving Abdominal Surgery Conditions: A Prospective Randomized Double-Blind Placebo Controlled Study
Brief Title: Pilot Study: Rectus Sheath Blocks for Improving Abdominal Surgery Conditions
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficult recruitment
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 203780
Record Dates: First submitted 2015-05-11; First posted 2015-05-19 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Hernia; Pain, Postoperative; Abdominal Wall Relaxation After Rectus Sheath Block
Keywords: Rectus Sheath Blocks; Abdominal Surgery
MeSH Terms: conditions — Hernia; Pain, Postoperative | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine (Active Comparator): Will have 20ml of bupivacaine injected into each rectus sheath.
  Interventions: Drug: Bupivacaine
- Normal Saline (Placebo Comparator): Will have 20ml of normal saline injected into each rectus sheath.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Bupivacaine — Using ultrasound guidance bupivacaine will be injected into the active group's rectus abdominis sheath.
  Other Names: Marcaine
  Arms: Bupivacaine
Drug: Normal Saline — Using ultrasound guidance normal saline will be injected into the placebo group's rectus abdominis sheath.
  Arms: Normal Saline

SUMMARY:
The purpose of this study is to show that the use of preoperative rectus sheath blocks can ultimately alleviate the need for using nondepolarizing muscle relaxants during certain abdominal procedures.

DETAILED DESCRIPTION:
The patients in the active group will be taken to the operating room and standard american society of anesthesiologists monitors will be applied. After induction of general anesthesia, the ultrasonographic anatomy of the umbilical region will be studied in each patient. The probe will be adjusted until optimum view of both rectus abdominis muscles, their sheaths and surrounding structures are identified. Once the umbilical region anatomy has been identified the puncture sites will be determined. The puncture sites will be aseptically prepped, the ultrasound probed will be covered with a sterile tegaderm, and sterile ultrasound gel will be used on the field. A 21-g EchoStim echogenic needle will be used. The needle will be inserted in the long axis parallel to the ultrasound probe. The needle will be advanced carefully until the needle tip is seen between the posterior aspect of the rectus muscle and its sheath. After a confirmed negative aspiration, 15 ml of 0.25% bupivacaine will be inserted in 2 ml increments, aspirating in between.

The placebo group will have the exact same procedure performed except 15 ml of normal saline will be injected in each rectus sheath instead of 0.25% bupivacaine. For all patients, when the block has been completed the surgery team will then prep the patient and proceed with the planned operation. The surgery staff and anesthesia providers taking care of the patient in the operating room will be unaware of the patient's group. At this point, all patients will be treated exactly the same. For intubation purposes, all patients will only receive succinylcholine. After intubation, elimination of the succinylcholine dose will be determined using a twitch monitor on the ulnar nerve. If at any point during the surgery, the surgery team needs more muscle relaxation then the anesthesia staff will give appropriate medications.

The first step will be to administer propofol 50mg IV, if hemodynamics allow, and to verify that the patient has 1.0-1.2 minimum alveolar concentration (MAC) of volatile anesthetic. If the patient is not at 1.0 MAC, then the volatile anesthetic should be increased. If this does not provide sufficient relaxation, then a nondepolarizing muscle relaxant will be given in 10mg increments titrated to a train of four of 2 twitches at the ulnar nerve. All patients will receive ofirmev and fentanyl in the operating room for pain control. Ofirmev 1000mg will be given pre-incision to each patient and 1.5 mcg/kg loading dose of fentanyl will be given to each patient. Fentanyl will be redosed in 50mcg increments for a 20% increase in blood pressure or heart rate above preinduction values that is sustained for 5 minutes despite an adequate depth of anesthesia, defined as 1 MAC or greater.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo an abdominal procedure with a periumbilical or midline incision above the umbilicus
* Age ≥ 18 years.
* American Society of Anesthesiologists physical status class 1 to 3

Exclusion Criteria:

* Known coagulopathy
* Preexisting muscular disease
* Medical conditions contraindicated to bupivacaine, succinylcholine or other medication used in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-01-01; Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Total consumption of nondepolarizing muscle relaxants used during abdominal surgery. | The duration of study therapy is only for the perioperative preparation period (usually 4-5 hrs) for the subject's abdominal procedure

CONTACTS AND LOCATIONS:
Overall Officials: Andrew G Cain, M.D., Principal Investigator — University of Arkansas
Locations (1):
- Univerisity of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Background] Kimura F, Oishi M, Yakoshi C, Ogasawara C, Ishihara H, Hirota K. [Rectus sheath block and transversus abdominis plane block for a patient with Lambert-Eaton myasthenic syndrome undergoing low anterior resection]. Masui. 2013 Aug;62(8):989-91. Japanese. PMID 23984583
- [Background] Quek KH, Phua DS. Bilateral rectus sheath blocks as the single anaesthetic technique for an open infraumbilical hernia repair. Singapore Med J. 2014 Mar;55(3):e39-41. doi: 10.11622/smedj.2014042. PMID 24664392
- [Background] Bashandy GM, Elkholy AH. Reducing postoperative opioid consumption by adding an ultrasound-guided rectus sheath block to multimodal analgesia for abdominal cancer surgery with midline incision. Anesth Pain Med. 2014 Aug 10;4(3):e18263. doi: 10.5812/aapm.18263. eCollection 2014 Aug. PMID 25289373